CLINICAL TRIAL: NCT01697826
Title: A Comparative Open Labeled Clinical Study to Evaluate the Efficacy and Tolerability of Two Different Intravaginal Formulations Containing a Combination of Clindamycin and Clotrimazole in Vaginal Infections
Brief Title: Comparison of Two Topical Formulations Containing Clindamycin and Clotrimazole in Patients With Vaginal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Bharti Daswani (Individual)
Collaborators: Resilient Cosmeceuticals Pvt. Ltd, Pune (Unknown)
Responsible Party: Sponsor-Investigator, Dr Bharti Daswani, Dr, Daswani, Bhart, M.D.
Organization: Daswani, Bhart, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ND1210132-34; CTRI/2011/04/001698 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2012-09-29; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Vaginal Infections
Keywords: Clindamycin; Clotrimazole; Vaginal formulation; Bacterial vaginosis; Candidiasis; Trichomoniasis; Mixed vaginitis; Infective vaginitis
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Candidiasis; Trichomonas Infections | interventions — Clindamycin; Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ClinSupV3 -soft gelatin capsule (Active Comparator): Soft gelatin capsule containing 100mg Clindamycin and 200mg clotrimazole administered per vaginally for 3 consecutive days
  Interventions: Drug: ClinSupV3 -soft gelatin capsule
- ClinSupV3ER- Extended release tablet (Active Comparator): ER tablets containing 100mg clindamycin and 200mg clotrimazole administered per vaginally for 3 consecutive days.
  Interventions: Drug: ClinSupV3ER- Extended release tablet

INTERVENTIONS:
Drug: ClinSupV3 -soft gelatin capsule — 3 day treatment with intravaginal formulation containing 100mg Clindamycin and 200mg clotrimazole
  Other Names: Clindamycin plus Clotrimazole
  Arms: ClinSupV3 -soft gelatin capsule
Drug: ClinSupV3ER- Extended release tablet — 3 day treatment with intravaginal formulation containing 100mg Clindamycin and 200mg Clotrimazole
  Other Names: Clindamycin plus Clotrimazole
  Arms: ClinSupV3ER- Extended release tablet

SUMMARY:
Randomized, Parallel Group, Active Controlled Trial to compare effectiveness and tolerability of 2 different vaginal formulations containing 200mg clotrimazole and clindamycin phosphate equivalent to 100mg clindamycin for 3 days in women clinically diagnosed to have infective vaginitis.

DETAILED DESCRIPTION:
* This is a Randomized, Comparative, Prospective, Open label, Single center study to compare the 3 day treatment course of intravaginal soft gelatin capsule containing clindamycin and clotrimazole versus intravaginal ER tablets of clindamycin and clotrimazole in patients with vaginal discharge and clinical diagnosis of bacterial, trichomonal, candidal or mixed vaginitis with respect to efficacy and tolerability; and to study the in vitro drug release pattern of intravaginal soft gelatin capsule and intravaginal ER tablets containing clindamycin and clotrimazole.
* The study will be conducted in B.J. Medical College & Sassoon General Hospitals, Pune. The study will be completed in 60 patients [30 patients in each group].
* The primary outcome measure is absence of any clinical sign suggestive of infective vaginitis and a vaginal swab that is negative for bacterial, trichomonal or candidal vaginitis at 8th day after start of treatment [Effectiveness in inducing a remission].
* The secondary outcome measures will be

  1. absence of any clinical sign suggestive of infective vaginitis and
  2. a vaginal swab that is negative for bacterial, trichomonal or candidal vaginitis at 29th day after start of treatment [Effectiveness in maintaining a remission] and ability to complete the 3day course without any break or experiencing intolerable side effects [Tolerability].

ELIGIBILITY:
Inclusion Criteria:

* Women with symptoms of vaginal discharge and/or odor and a clinical diagnosis of vaginitis of infective origin [based on symptoms and signs on per speculum examination]
* Age at least 18 years
* Capable of giving written informed consent
* Agree to no intercourse for 8 days from the day of start of treatment
* Agree not to douche or use any intravaginal products during the study period (including tampons, medications and devices)

Exclusion Criteria:

* Post-menopausal women
* Menstruating at diagnosis
* Pregnancy
* Any antifungal or antibiotic use 14 days prior to enrolment
* Use of oral or intravaginal antibiotics within the past 2 weeks
* Immunosuppressive drug within 4 months
* Presence of vaginal / vulval ulcer
* Presence of any other vulval, vaginal or medical condition, including cervical neoplasia/ treatment that might confound treatment response
* Inability to keep return appointments
* History of hypersensitivity to clotrimazole, clindamycin or lincomycin
* History of regional enteritis, ulcerative colitis or antibiotic associated colitis
* Significant disease or acute illness that in the Investigators assessment could complicate the evaluation
* Intrauterine Device

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure for Global effectiveness | On 8th day after start of treatment
  Number of patients showing resolution of clinical signs suggestive of infective vaginitis and a vaginal swab that is negative for bacterial, trichomonal or candidal vaginitis

SECONDARY OUTCOMES:
Secondary outcome measures for Global effectiveness | 29th day after initiation of treatment
  Number of patients showing absence of clinical signs suggestive of infective vaginitis and a vaginal swab that is negative for bacterial,trichomonal or candidal vaginitis
Secondary outcome measures for tolerability | 8th day after start of treatment
  Number of patients that are able to successfully complete the 3 day treatment course without a break or experiencing intolerable side-effects

OTHER OUTCOMES:
Clinical Response | at 8th day and 29th day after initiation of treatment
  Number of the patients showing normalization of vaginal pH to 4.5
Clinical response | at 8th and 29th day after start of treatment
  Number of the patients achieving improvement in scores for quantity of vaginal discharge by at least 1 unit from baseline
Clinical response | at 8th day and 29th day after start of treatment
  Number of the patients achieving improvement in scores for itching by at least 1 unit from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bharti R Daswani, MD, PhD, Principal Investigator — BJ Govt Medical College & Sassoon General Hospitals, Pune
Locations (1):
- BJ Govt. Medical College & Sassoon General Hospitals, Pune, Pune, Maharashtra, India